CLINICAL TRIAL: NCT06825481
Title: Uterine Doppler As StillbirthPredictor
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: StUtDop1.0
Record Dates: First submitted 2024-12-30; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-10

CONDITIONS: Intrauterine Fetal Death
Keywords: Uterine Doppler
MeSH Terms: conditions — Stillbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to define the predictive value of intrauterine fetal death for different longitudinal patterns of uterine artery Doppler indices (UtA-PI, UtA-RI and notch) from the second and third trimester of pregnancy in patients admitted with a diagnosis of intrauterine foetal death in the period January 2010-April 2020.

DETAILED DESCRIPTION:
No changes in the obstetrical conduct of patients with MEFs are expected, since the data will be analysed retrospectively in patients in whom the event of intrauterine foetal death has already occurred. Patients will be treated according to normal clinical protocols.

The following information will be recorded for each patient

* Age
* Body mass index (BMI)
* Ethnicity
* Parity
* Method of pregnancy onset (spontaneous vs. medically assisted procreation)
* Maternal pathologies (if any)
* Any foetal pathologies
* Ultrasound parameters in the second and third trimester of pregnancy

  * Estimation of fetal weight
  * Umbilical artery Doppler (UA-PI)
  * Uterine artery Doppler (UtA-PI, UtA-RI and notch)
* Gestational age of fetal endouterine death
* Type of delivery
* Newborn and placental weight
* Histopathological findings of newborn and annexes (placenta and umbilical cord)

ELIGIBILITY:
Inclusion Criteria:

* Fetal endouterine death in single pregnancies with gestation period ≥ 24 weeks
* Obtaining informed consent form

Exclusion Criteria:

* Multiple pregnancies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Assuming a standard deviation of 0.5 in the Doppler values of both cases and controls and a difference in the intercepts of 30% of the two regression lines, it is estimated that 72 cases and 4791 controls are needed to obtain a power of 80% at a type I error of 5%. The controls will be represented by the Doppler values reported in the literature for pregnancies not complicated by MEF.
Sampling Method: Non-Probability Sample
Enrollment: 4863 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the association between uterine artery Doppler indexes (UtA-PI, UtA-RI and notch) and MEF | From the 13th to the 24th weeks of pregnancy
  Data will be analyzed by routine univariate descriptive analysis. Doppler values, which represent the main predictive parameter of study in order to find a possible association with the outcome of interest, will be analyzed longitudinally by means of a mixed linear model, a multivariate model capable of evaluating at the same time both the values of the exploratory variable of interest (Doppler) and possible covariates.
  In addition, the mixed model is also capable of evaluating the "individual-specific" or random effect, the purpose of which is to isolate as precisely as possible the effect due to the variable hypothesized to be predictive toward the outcome of interest. In order to evaluate the hypothetically aberrant Doppler value compared to the expected normal value, a physiological control population will be recruited for both outcome and Doppler values.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Farina, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy